CLINICAL TRIAL: NCT04154930
Title: A Randomized, Evaluator-blinded, Parallel Group, No-treatment Controlled, Multi-center Study to Evaluate the Safety and Effectiveness of Restylane-L® for Correction of Infraorbital Hollows
Brief Title: Restylane-L for Correction of Infraorbital Hollows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USTT1904
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Results first posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Infraorbital Hollows
Keywords: Tear Trough

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Restylane-L Treatment (Experimental): Restylane-L® injected with optional touch-up at 1 month and optional retreatment at 12 months.
  Interventions: Device: Restylane-L®
- No Treatment Control (No Intervention): No treatment control with optional treatment at 12 months.

INTERVENTIONS:
Device: Restylane-L® — Intradermal injection.
  Arms: Restylane-L Treatment

SUMMARY:
This is a prospective, randomized, evaluator-blinded, no-treatment controlled, parallel group, multi-center US study to evaluate the safety and effectiveness of Restylane-L® for correction of Infraorbital Hollows.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe infraorbital hollows with no more than one grade difference between the left and right side at baseline as assessed by the blinded evaluator.
* Males or non-pregnant, non-breastfeeding females, over the age of 21.
* Intent to undergo correction of both orbital hollows.

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel or to gram positive bacterial proteins.
* Known/previous allergy or hypersensitivity to local anesthetics, e.g. lidocaine or other amide-type anesthetics.
* Previous deep and/or superficial facial dermal therapies.
* Active or a history of recurrent or chronic infraorbital edema or rosacea or uncontrolled severe seasonal allergies.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Galderma Research Site, Encino, California
  - Galderma Research Site, Los Angeles, California
  - Galderma Research Site, Redondo Beach, California
  - Galderma Research Site, Solana Beach, California
  - Galderma Research Site, Westport, Connecticut
  - Galderma Research Site, Boynton Beach, Florida
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, West Palm Beach, Florida
  - Galderma Research Site, Chicago, Illinois
  - Galderma Research Site, Chestnut Hill, Massachusetts
  - Galderma Research Site, New York, New York
  - Galderma Research Site, Rochester, New York
  - Galderma Research Site, Wilmington, North Carolina
  - Galderma Research Site, Nashville, Tennessee
  - Galderma Research Site, Spring, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 sites in the United States from 11 November 2019 to 06 April 2022.
Groups:
- Restylane-L® Treatment: Participants were injected with Restylane-L® intradermal injection using either needle or cannula on Day 1, optional touch-up injection administered at 1 month of initial treatment.
- No Treatment Control: No-treatment control group did not receive any treatment during the main study period.
Period: Overall Study
Arm/Group | Restylane-L® Treatment | No Treatment Control
Started | 287 | 46
Completed | 250 | 33
Not Completed | 37 | 13
Not completed — Withdrawal by Subject | 15 | 6
Not completed — Withdrew consent- Covid-19 related | 2 | 1
Not completed — Lost to Follow-up | 14 | 6
Not completed — Other | 6 | 0

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population included all participants who were randomized at baseline and analyzed according to the randomization scheme determined at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane-L® Treatment | No Treatment Control | Total
Number analyzed (Participants) | 287 | 46 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (11.58) | 45.5 (12.27) | 44.4 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 38 | 290
  Male | 35 | 8 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66 | 9 | 75
  Not Hispanic or Latino | 221 | 37 | 258
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White: White | 257 | 39 | 296
  White: Black or African American | 17 | 4 | 21
  White: Asian | 4 | 1 | 5
  White: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White: Other | 8 | 2 | 10
Fitzpatrick skin type (FST) [Count of Participants; unit: Participants] — FST I: white; very fair; red or blond hair; blue eyes; freckles. always burns, never tans.
  FST II: white; fair; red or blond hair; blue, hazel or green eyes. usually burns, tans with difficulty.
  FST III: cream white; fair with any eye or hair color; very common. sometimes mild burn, gradually tans.
  FST IV: brown; typical Mediterranean Caucasian skin. rarely burns, tans with ease.
  FST V: dark brown; Middle Eastern skin types. very rarely burns, tans very easily.
  FST VI: Skin color - black. Skin Characteristics - never burns, tans very easily.
  Participants
    FST I | 5 | 0 | 5
    FST II | 75 | 11 | 86
    FST III | 117 | 20 | 137
    FST IV | 62 | 10 | 72
    FST V | 13 | 3 | 16
    FST VI | 15 | 2 | 17
Blinded Evaluator GIHS score - left [Count of Participants; unit: Participants] — Galderma Infraorbital Hollows Scale (GIHS) is a validated 4-point scale used to assess Infraorbital Hollows: 0 (none [hollowness]),1 (mild [hollowness]), 2 (moderate [hollowness]), 3 (severe [hollowness])
  Participants
    0 | 0 | 0 | 0
    1 | 0 | 0 | 0
    2 | 147 | 27 | 174
    3 | 140 | 19 | 159
Blinded Evaluator GIHS score - right [Count of Participants; unit: Participants] — Galderma Infraorbital Hollows Scale (GIHS) is a validated 4-point scale used to assess Infraorbital Hollows: 0 (none [hollowness]),1 (mild [hollowness]), 2 (moderate [hollowness]), 3 (severe [hollowness])
  Participants
    0 | 0 | 0 | 0
    1 | 0 | 0 | 0
    2 | 147 | 24 | 171
    3 | 140 | 22 | 162

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate Based on the Blinded Evaluator's Live Assessment of the Galderma Infraorbital Hollows Scale (GIHS)
Description: Responder rate was defined as the percentage of participants with at least a 1-point improvement from baseline on the Galderma Infraorbital Hollows Scale (GIHS), on both sides of the face, concurrently. GIHS is a validated 4-point scale used to assess Infraorbital Hollows: 0 (none [hollowness]), 1 (mild [hollowness]), 2 (moderate [hollowness]), 3 (severe [hollowness]). Higher score means more severe (worse) hollowness in the infraorbital Hollows.
Time Frame: At 3 months after Baseline
Population: The modified intention-to-treat (mITT) population included all participants who were randomized and analyzed according to the randomization scheme and who did not have a GIHS Month 3 visit assessment conducted remotely (i.e., remote study visit and/or GIHS assessment performed remotely).
Measure: Number; unit: Percentage of participants
Arm/Group | Restylane-L® Treatment | No Treatment Control
Number analyzed (Participants) | 210 | 35
Percentage of participants | 87.4 | 17.7
Statistical Analysis 1: Comparison: Restylane-L® Treatment vs No Treatment Control; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Treatment difference = 69.7, 95% CI 2-sided [52.54 to 86.89]

2. Secondary Outcome: Responder Rate Based on the Blinded Evaluator's Live Assessment of the GIHS at 6, 9, and 12 Months After Baseline And at 3 and 6 Months After Optional Treatment
Description: Responder rate was defined as the percentage of participants with at least a 1-point improvement from baseline on the GIHS, on both sides of the face, concurrently at each of the timepoints. GIHS is a validated 4-point scale used to assess Infraorbital Hollows: 0 (none [hollowness]), 1 (mild [hollowness]), 2 (moderate [hollowness]), 3 (severe [hollowness]). Higher score means more severe (worse) hollowness in the infraorbital Hollows.
Time Frame: At 6, 9, and 12 months after Baseline and at 3 and 6 months after optional treatment
Population: mITT population included all participants who were randomized and analyzed according to the randomization scheme and who did not have a GIHS Month 3 visit assessment conducted remotely (that is [i.e.], remote study visits and/or GIHS assessment performed remotely). Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Restylane-L® Treatment | No Treatment Control
Number analyzed (Participants) | 257 | 37
Percentage of participants
  At Month 6 | 86.0 | 13.5
  At Month 9: number analyzed (Participants) | 254 | 36
  At Month 9 | 77.6 | 11.1
  At Month 12: number analyzed (Participants) | 255 | 36
  At Month 12 | 63.5 | 11.1
  At Month 3 after optional treatment: number analyzed (Participants) | 155 | 29
  At Month 3 after optional treatment | 87.1 | 82.8
  At Month 6 after optional treatment: number analyzed (Participants) | 157 | 29
  At Month 6 after optional treatment | 80.3 | 65.5
Statistical Analysis 1: Comparison: Restylane-L® Treatment vs No Treatment Control; Responder Rate Based on the Blinded Evaluator's live assessment of the GIHS at 6 Months After Baseline; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Treatment difference = 72.5, 95% CI 2-sided [60.67 to 84.28]
Statistical Analysis 2: Comparison: Restylane-L® Treatment vs No Treatment Control; Responder Rate Based on the Blinded Evaluator's live assessment of the GIHS at 9 Months After Baseline; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Treatment difference = 66.4, 95% CI 2-sided [54.97 to 77.92]
Statistical Analysis 3: Comparison: Restylane-L® Treatment vs No Treatment Control; Responder Rate Based on the Blinded Evaluator's live assessment of the GIHS at 12 Months After Baseline; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Treatment difference = 52.4, 95% CI 2-sided [40.57 to 64.26]

3. Secondary Outcome: Percentage of Participants With At Least "Improved" on the Global Aesthetic Improvement Scale (GAIS) Based on the Participants Live Assessment
Description: GAIS responder rates are based on independent assessments by the participant. Responder rate was defined as the percentage of participants with at least "Improved" when compared to baseline before first treatment. The 7-graded GAIS was used by the participant to live assess the aesthetic improvement of the infraorbital hollows by responding to the question: "How would you describe the aesthetic improvement of your tear troughs today compared to the photograph taken before treatment?" by using the respective categorical scale as follows; Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse.
Time Frame: At 1, 3, 6, 9, and 12 months after randomization, at 1 month after optional touch-up, and at 1, 3 and 6 months after optional treatment
Population: ITT population included all participants who were randomized and analyzed according to the randomization scheme. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Restylane-L® Treatment | No Treatment Control
Number analyzed (Participants) | 272 | 38
Percentage of participants
  At Month 1: number analyzed (Participants) | 272 | 35
  At Month 1 | 93.0 | 2.9
  At Month 3: number analyzed (Participants) | 258 | 38
  At Month 3 | 95.0 | 2.6
  At Month 6: number analyzed (Participants) | 257 | 37
  At Month 6 | 91.8 | 0
  At Month 9: number analyzed (Participants) | 253 | 36
  At Month 9 | 88.1 | 0
  At Month 12: number analyzed (Participants) | 257 | 36
  At Month 12 | 79.8 | 2.8
  At Month 1 after optional touch up: number analyzed (Participants) | 198 | 0
  At Month 1 after optional touch up | 99.0 |
  At Month 1 after optional treatment: number analyzed (Participants) | 155 | 32
  At Month 1 after optional treatment | 98.7 | 93.8
  At Month 3 after optional treatment: number analyzed (Participants) | 157 | 29
  At Month 3 after optional treatment | 94.3 | 89.7
  At Month 6 after optional treatment: number analyzed (Participants) | 158 | 29
  At Month 6 after optional treatment | 93.0 | 82.8

4. Secondary Outcome: Percentage of Participants With At Least "Improved" on the GAIS Based on the Treating Investigator Live Assessment
Description: GAIS responder rates are based on independent assessments by the Treating Investigator. Responder rate was defined as the percentage of participants with at least "Improved" when compared to baseline before first treatment. The 7-graded GAIS was used by the treating investigator to live assess the aesthetic improvement of the infraorbital hollows by responding to the question: "How would you describe the aesthetic improvement of participant's tear troughs today compared to the photograph taken before treatment?" by using the respective categorical scale as follows; Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Restylane-L® Treatment | No Treatment Control
Number analyzed (Participants) | 271 | 39
Percentage of participants
  At Month 1: number analyzed (Participants) | 271 | 35
  At Month 1 | 97.4 | 2.9
  At Month 3: number analyzed (Participants) | 257 | 39
  At Month 3 | 97.7 | 5.1
  At Month 6: number analyzed (Participants) | 257 | 37
  At Month 6 | 95.3 | 10.8
  At Month 9: number analyzed (Participants) | 255 | 36
  At Month 9 | 92.5 | 5.6
  At Month 12: number analyzed (Participants) | 257 | 36
  At Month 12 | 87.5 | 2.8
  At Month 1 after optional touch up: number analyzed (Participants) | 199 | 0
  At Month 1 after optional touch up | 99.5 |
  At Month 1 after optional treatment: number analyzed (Participants) | 155 | 32
  At Month 1 after optional treatment | 100 | 100
  At Month 3 after optional treatment: number analyzed (Participants) | 156 | 29
  At Month 3 after optional treatment | 97.4 | 96.6
  At Month 6 after optional treatment: number analyzed (Participants) | 158 | 29
  At Month 6 after optional treatment | 99.4 | 89.7

ADVERSE EVENTS:
Time Frame: From randomization up to 18 months
Description: Safety population includes all subjects who were treated with Restylane-L or randomized to the control group
Arm/Group | Restylane-L® Treatment | No Treatment Control
All-Cause Mortality (participants affected / at risk) | 1/287 | 0/46
Serious Adverse Events (participants affected / at risk) | 4/287 | 0/46
Other Adverse Events (participants affected / at risk) | 97/287 | 6/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane-L® Treatment (N=287) | No Treatment Control (N=46)
COVID 19 (Infections and infestations) | 2 (2) | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane-L® Treatment (N=287) | No Treatment Control (N=46)
Migraine (Nervous system disorders) | 3 (3) | 1 (1)
COVID 19 (Infections and infestations) | 15 (15) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 30 (30) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (8) | 0 (0)
Hordeolum (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 0 (0) — Common Cold
Diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bipolar Disorder II (Psychiatric disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) — Numbness
COVID 19 Vaccine reaction (Immune system disorders) | 4 (11) | 0 (0) — fever, body ache, rash, swelling, migraine, chills, headache
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomachache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Immune system disorders) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Herniated disk (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spontaneous Breast Implant Rupture (Product Issues) | 1 (1) | 0 (0)
ADHD (Psychiatric disorders) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Nervous system disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysplastic naevus (Eye disorders) | 1 (1) | 0 (0)
acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
polycystic ovary syndrome (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Lupus erythematosus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Viral rhinitis (Infections and infestations) | 2 (2) | 0 (0)
Injury due to fall (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Strep throat (Infections and infestations) | 1 (1) | 0 (0)
Vulval abcess (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Binge drinking (Psychiatric disorders) | 1 (1) | 0 (0)
Benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Benign mass in right breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Autoimmune Disorder (Immune system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0)
Implant Site Swelling (General disorders) | 12 (26) | 0 (0)
Implant Site Pain (General disorders) | 8 (13) | 0 (0)
Implant Site Bruising (General disorders) | 5 (7) | 0 (0)
Implant Site Mass (General disorders) | 4 (4) | 0 (0)
Implant Site Oedema (General disorders) | 4 (7) | 0 (0)
Implant Site Pruritus (General disorders) | 2 (2) | 0 (0)
Implant Site Discolouration (General disorders) | 1 (1) | 0 (0)
Skin Discolouration (General disorders) | 2 (2) | 0 (0)
Implant Site Induration (General disorders) | 1 (1) | 0 (0)
Implant Site Paraesthesia (General disorders) | 1 (1) | 0 (0)
Post Inflammatory Pigmentation Change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Dryness (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04154930/Prot_004.pdf
  • Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT04154930/SAP_005.pdf